CLINICAL TRIAL: NCT03015649
Title: Evaluation of Longer Duration Use of the SAVI SCOUT Surgical Guidance System for Excision of Breast and Axillary Lesions in Neo-adjuvant Therapy Patients: A Pilot Study
Brief Title: Long Term Use of SAVI SCOUT: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envision Healthcare Scientific Intelligence, Inc. (Other)
Collaborators: Cianna Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CMI-SCOUT-001
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Breast Diseases
Keywords: breast cancer; neoadjuvant treatment; surgical guidance system
MeSH Terms: conditions — Breast Diseases; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCOUT device (Experimental): The study population consists of 25 - 35 adult surgical patient volunteers who plan to have definitive breast cancer surgery at Memorial Healthcare System (MHS) Hospitals after neoadjuvant treatment.
  The investigator will identify subjects who meet inclusion/exclusion criteria, obtain patient's consent and schedule the subject for the SAVI SCOUT Surgical Guidance System procedure. All study participants will receive the same treatment assignment, i.e. lesion localization with the SCOUT device 31 - 365 days prior to surgery. Neoadjuvant treatment decisions will be determined by patient's medical oncologist.
  Interventions: Device: SAVI SCOUT Surgical Guidance System

INTERVENTIONS:
Device: SAVI SCOUT Surgical Guidance System — SAVI SCOUT Surgical Guidance System is a non-wire system, which uses nonradioactive light-activated radar, to provide breast surgeons with real-time guidance to locate and remove the target lesion in the breast and/or axillary tissue.

SUMMARY:
The purpose of this study is to evaluate the performance of FDA-cleared SAVI SCOUT Breast Localization and Surgical Guidance System (SCOUT) over a longer duration prior to surgery. The device is a non-wire system, which uses nonradioactive light-activated radar, to provide breast surgeons with real-time guidance to locate and remove the target lesion in the breast and/or axillary tissue. The SCOUT device standard of care use is placement up to 30 days prior to surgery to assist surgeons in the localization and retrieval of breast/axillary lesions. Routine image-guided methods (Mammography, Ultrasound, and CT) are used. In this study, investigators will assess the longer term placement of the SCOUT device over an extended time (31 - 365 days) in order to address the needs of patients who require neoadjuvant treatment prior to definitive surgery.

DETAILED DESCRIPTION:
The SAVI SCOUT (Cianna Medical, Inc.) surgical guidance system received 510(k) U.S. Food and Drug Administration (FDA) approval in August 2014. This system is used as a standard of care since 2015 in the Memorial Healthcare System (MHS) operating rooms by experienced breast surgeons (over 150 MHS breast cancer patients and over 5,000 U.S. breast cancer patients as of September 2016). In MHS standard of care practice, the device is placed at the target lesion(s) under image-guidance by the radiologist up to 30 days prior to surgery.

Patients with certain types of breast cancer undergo neoadjuvant treatment with biologic (hormonal) and/or chemotherapy with the goal of decreasing the tumor volume prior to definitive surgery. If the original cancer lesion(s) resolve completely, this is called complete pathologic response (pCR). pCR and even a partial response, while good for the patient, can result in disappearance or poor visualization of the target and often render pre-operative image-guided localization by the radiologist more difficult and less reliable. This can result in unintended larger, more disfiguring breast cancer surgery. Therefore, if the SCOUT device can be placed prior to treatment response, when the lesion is clearly visualized on imaging, accurate image-guided targeting is optimal and thus placement and subsequent surgery should be more accurate. If this pilot study demonstrates successful performance of the device without device-related complications, it will bring improved value to future patients who will require fewer and/or less extensive pre-operative and surgical procedures. Some value may also be provided to subjects as the targeting before tumor shrinkage is expected to be more accurate.

Thus, this pilot study will assess the performance of FDA-cleared SCOUT system over a longer duration prior to breast and/or axillary lymph node surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide informed consent. Patient SCOUT device(s) is placed as part of routine care or study but before neoadjuvant treatment begins.
* Patient is female.
* Patient is between the ages of 18 and 90 years.
* Patient has breast cancer and will undergo neoadjuvant therapy and excision at Memorial Healthcare System.
* Patient is willing and able to comply with all study procedures and be available to follow-up for the duration of the study (1 - 13 months).
* Patient reads or understands English or Spanish.

Exclusion Criteria:

* Patient is pregnant.
* Patient has pacemaker or implantable defibrillators (These have not been bench tested as of September 2016).
* Patient has known or suspected nickel allergy.
* Patient is scheduled or receiving investigational drugs for neoadjuvant regimen. (This could confound UADE of this device.)
* Patient has any condition that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
* Patient has other malignancy except for adequately treated and cured basal or squamous cancer, curatively treated in situ disease or any other cancer for which the patient has been disease free for greater than or equal to 5 years.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hayes-Macaluso, MD, Principal Investigator — Envision Healthcare Scientific Intelligence, Inc.
Locations (1):
- Envision Physician Scientific Research, Inc. formerly Sheridan Healthcare, Inc., Plantation, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox CE, Garcia-Henriquez N, Glancy MJ, Whitworth P, Cox JM, Themar-Geck M, Prati R, Jung M, Russell S, Appleton K, King J, Shivers SC. Pilot Study of a New Nonradioactive Surgical Guidance Technology for Locating Nonpalpable Breast Lesions. Ann Surg Oncol. 2016 Jun;23(6):1824-30. doi: 10.1245/s10434-015-5079-x. Epub 2016 Feb 3. PMID 26847680
- [Background] Caudle AS, Yang WT, Mittendorf EA, Black DM, Hwang R, Hobbs B, Hunt KK, Krishnamurthy S, Kuerer HM. Selective surgical localization of axillary lymph nodes containing metastases in patients with breast cancer: a prospective feasibility trial. JAMA Surg. 2015 Feb;150(2):137-43. doi: 10.1001/jamasurg.2014.1086. PMID 25517573
- [Background] Hylton NM, Gatsonis CA, Rosen MA, Lehman CD, Newitt DC, Partridge SC, Bernreuter WK, Pisano ED, Morris EA, Weatherall PT, Polin SM, Newstead GM, Marques HS, Esserman LJ, Schnall MD; ACRIN 6657 Trial Team and I-SPY 1 TRIAL Investigators. Neoadjuvant Chemotherapy for Breast Cancer: Functional Tumor Volume by MR Imaging Predicts Recurrence-free Survival-Results from the ACRIN 6657/CALGB 150007 I-SPY 1 TRIAL. Radiology. 2016 Apr;279(1):44-55. doi: 10.1148/radiol.2015150013. Epub 2015 Dec 1. PMID 26624971
- [Background] Mango V, Ha R, Gomberawalla A, Wynn R, Feldman S. Evaluation of the SAVI SCOUT Surgical Guidance System for Localization and Excision of Nonpalpable Breast Lesions: A Feasibility Study. AJR Am J Roentgenol. 2016 Oct;207(4):W69-W72. doi: 10.2214/AJR.15.15962. Epub 2016 Jun 15. PMID 27304083

RESULTS

PARTICIPANT FLOW:
Groups:
- SCOUT Device: All study participants received the same treatment assignment, i.e. lesion localization with the SCOUT device 31 - 365 days prior to surgery. Each participant underwent the SAVI SCOUT Surgical Guidance System procedure.
Period: Overall Study
Arm/Group | SCOUT Device
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SCOUT Device
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 50 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  African American | 12
  Hispanic | 11
  Other | 1
Node Positive [Count of Participants; unit: Participants] | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Considered to Have a Successful Surgery
Description: The primary endpoint of this study is successful surgery. Successful surgery (defined as one where the device stays in place and can be removed successfully during surgery) when this device is placed 31 - 365 days prior to surgery. Unsuccessful surgery is defined as one where the device does not stay in place and/or cannot be removed successfully during surgery) when this device is placed 31 - 365 days prior to surgery.
Time Frame: 31 - 365 days prior to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | SCOUT Device
Number analyzed (Participants) | 34
Participants | 34

ADVERSE EVENTS:
Time Frame: 0 months - 14 months. Reportable adverse events were collected from the time after informed consent is obtained until 30 days (for non-serious AEs) or 7 days (for SAEs) after the last day of study participation
Description: Adverse events from underlying diseases and related to neoadjuvant treatments were not intended to be collected. The written Protocol was amended to clarify this point. All reported SAEs were unrelated to the investigational device and collected prior to the Protocol amendment. The collected events were all previously known as anticipated side effects of chemotherapy and fertility preservation.
Arm/Group | SCOUT Device
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

LIMITATIONS AND CAVEATS:
Principal Investigator has left the organization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03015649/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03015649/Prot_SAP_001.pdf